CLINICAL TRIAL: NCT03132025
Title: Phase 1 Study of Apatinib and Capecitabine Combination to Maintain Treating Metastatic Colorectal Cancer
Brief Title: Study of Apatinib and Capecitabine Combination to Maintain Treating Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqiao Zhang (Other)
Responsible Party: Sponsor-Investigator, Yanqiao Zhang, Head of Gastroenterology, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 045186298222
Record Dates: First submitted 2017-03-16; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Apatinib; Capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib; Capecitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: "apatinib" and "capecitabine" (Experimental): Arm A: "apatinib" and "capecitabine" apatinib 250mg qdpo; capecitabine 1000mg/m2 qdpo d1-14 q3w
  Interventions: Drug: "Apatinib" and "Capecitabine"
- B: "capecitabine" single drug (Active Comparator): Arm B: "capecitabine" single drug "capecitabine" 1000mg/m2 qdpo d1-14 q3w
  Interventions: Drug: "Capecitabine"

INTERVENTIONS:
Drug: "Apatinib" and "Capecitabine" — Combine "Apatinib" and "Capecitabine" to Maintain Treating Metastatic Colorectal Cancer
  Other Names: Arm A
  Arms: A: "apatinib" and "capecitabine"
Drug: "Capecitabine" — Single Drug "Capecitabine" to Maintain Treating Metastatic Colorectal Cancer
  Other Names: Arm B
  Arms: B: "capecitabine" single drug

SUMMARY:
To control apatinib and capecitabine combination to maintain treating metastatic colorectal cancer.

DETAILED DESCRIPTION:
To control apatinib and capecitabine combination to maintain treating metastatic colorectal cancer,primary endpoint include in mPFS; secondary endpoint include in mOS, tolerance and security.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form should be issued prior to conducting any research process;
2. Men or women aged 18-75 years;
3. Patients with advanced and / or metastatic colorectal cancer confirmed by histology or cytology;
4. Patients who has not exposed to apatinib previously and had received oxaliplatin combined with fluorouracil chemotherapy;
5. The estimated survival time is longer than 3 months;
6. ECOG score was 0 or 1;
7. According to the RECIST v1.1 guidance, at least 1 lesion(who had not received radiotherapy) showed that the longest diameter≥10mm(except for lymph node, the short axis of the lymph node must be≥15mm) through CT or MRI(intravenous contrast agent was preferred ) accurate measurement and the lesion should be suitable for repeatable and accurate measurement; the lesion located in the previously irradiated area can be used as a measurable lesion if the lesion was proved in progress;
8. With sufficient organ and bone marrow function, defined as follows:

   * Hb≥9 g/dL
   * Absolute neutrophil count ≥1.0 × 109 /L
   * Platelet count≥75 × 109 /L
   * Serum bilirubin ≤ 1.5 × ULN, which would not be appropriate for patients with Gilbert syndrome (Persistent or recurrent hyperbilirubinemia, mainly unconjugated bilirubin, with no evidence of hemolysis or abnormal liver pathology) which can consult a doctor
   * ALT&AST ≤ 2.5 × ULN; for patients with liver metastases, ALT&AST ≤ 5 × ULN Calculate the creatinine clearance rate by Cockcroft-Gault formula
   * Creatinine clearance rate measured( by actual body weight) or by measuring urine collection for 24 hours> 40 mL/min(the value of the measurement of the 24 - hour urine collection will be used to determine eligibility if the two methods are used)
9. Women of childbearing age must have a pregnancy test (serum or urine) within 7 days before inclusion, the results should be negative and they are willing to use the appropriate methods of contraception during the trial and within 6 months of the last experimental drug administration. Men should agree to use appropriate methods of contraception during the trial and within 6 months of the last experimental drug administration;
10. Patients volunteered to participate in the trial and signed informed consent form with good compliance.

Exclusion Criteria:

1. Patients with hypertension and can not be reduced to the normal range with antihypertensive drugs(systolic pressure >140 mmHg / diastolic pressure > 90 mmHg),patients with coronary heart disease more than grade II, arrhythmia (including QTc interval Prolongation men>450 ms, women >470 ms) and cardiac insufficiency;
2. With a variety of factors affecting oral drugs(such as unable to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction, etc.);
3. Special note: patients with the risk of gastrointestinal bleeding can not be included, including the following: active peptic ulcer lesions and fecal occult blood (+ +); patients with melena and hematemesis in 3 months; for patients with fecal occult blood (+) and primary gastric tumor without surgery should be carried out gastroscopy, patients with ulcero carcinoma of stomach and believed to cause the lesion to bleed by the physician;
4. Abnormal coagulation function(INR>1.5×ULN、 APTT>1.5×ULN) with bleeding tendency;
5. With Symptomatic central nervous system metastasis;
6. Pregnant or lactating women;
7. Other patients unsuitable for inclusion considered by the physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-30 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival of Patients with Apatinib and Capecitabine Combination That is prolonged | up to 10 months
  Patients with double drug group have more longer progression-free survival (PFS) than patients with single drug group

IPD SHARING:
Plan to Share IPD: Undecided